CLINICAL TRIAL: NCT00844662
Title: An Open, Randomised, Controlled, Parallel Group, Phase III Study to Investigate the Safety and Efficacy of Fermagate and Sevelamer Hydrochloride in Haemodialysis Patients With Hyperphosphataemia
Brief Title: Phase III Study to Investigate the Safety and Efficacy of Fermagate and Sevelamer Hydrochloride
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Ineos Healthcare Limited (Industry)
Responsible Party: Study Project Manager, INEOS Healthcare Limited
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT 402; 2008-004730-25 (EudraCT Number)
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2010-10-19 (Estimated); Status verified 2010-10

CONDITIONS: Chronic Kidney Failure
Keywords: Hyperphosphataemia; phosphate binder
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperphosphatemia | interventions — iron-magnesium hydroxycarbonate; Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Fermagate
- 2 (Active Comparator)
  Interventions: Drug: Sevelamer hydrochloride

INTERVENTIONS:
Drug: Fermagate — Film coated tablet 500mg
  Other Names: Alpharen
  Arms: 1
Drug: Sevelamer hydrochloride — Tablet 800mg
  Other Names: Renagel
  Arms: 2

SUMMARY:
Magnesium iron hydroxycarbonate is a phosphate binder that absorbs phosphate from food, reducing the amount that the body can absorb.

The purpose of this study is to assess the efficacy of magnesium iron hydroxycarbonate in subjects requiring haemodialysis, compared with a marketed phosphate binder, sevelamer hydrochloride.

DETAILED DESCRIPTION:
High levels of phosphate in the blood are linked with serious effects, due to calcium imbalances (high levels of parathyroid hormone (PTH), bone disease, formation of calcium deposites in the body and blood-vessel disease.

Current guidelines indicate that blood phosphorous levels should be maintained between 1.13 to 1.78mmol/L in patients who receive haemodialysis.

The purpose of this study is to establish the non-inferiority of magnesium iron hydroxycarbonate to sevelamer hydrochloride in lowering serum phosphate in haemodialysis patients treated for 3 months. Additional objectives: (1) to determine the safety of magnesium iron hydroxycarbonate after short term (3 months) and long term (6 and 12 months) treatment, (2)to determine the efficacy of magnesium iron hydroxycarbonate after long term treatment (6 and 12 months) and (3) To compare the effects of magnesium iron hydroxycarbonate and sevelamer hydrochloride on measures of mineral metabolism, albumin, pre-albumin and iron status after short term (3 months) and long term (6 and 12 months) treatment.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be considered eligible for entry in the study if they meet all of the following criteria.

1. Male or female, aged > 18 years.
2. Able to comply with the study procedures and medication.
3. Written informed consent given.
4. On a stable haemodialysis regimen (at least 3x per week) for ≥12 weeks prior to screening.
5. (a) Subject receiving phosphate binder medication(s) at screening, must have been on a stable regimen (dose and medication) for at least 1 month prior to screening and will remain on this regimen until entry into the washout period OR (b)Subject (i) is not currently receiving any phosphate binding medication at screening (or medication likely to act as a phosphate binder) and (ii) must not have done so for at least one month and (iii) has sustained hyperphosphataemia.
6. Willing to abstain from taking any phosphate binder or oral magnesium-, oral aluminium- or oral iron-containing products and preparations other than the study medication.
7. If required to take >6000 mg/day of fermagate, the subject will be willing to have at least three meals per day.

   Specifically, for randomisation and inclusion into the treatment period, the following criterion must be fulfilled:
8. Has a serum phosphate value of ≥1.94 mmol/L (≥6.0 mg/dL) within the 2 to 4 week washout period or above 3.0 mmol/L (9.3 mg/dL) at any time during washout.

Exclusion Criteria:

Subjects will not be considered eligible for entry in the study if they meet one or more of the following criteria.

1. Participation in any clinical trial using an investigational product or device during the 30 days preceding the Screening Visit.
2. Previous experience of fermagate treatment.
3. A significant history of alcohol, drug or solvent abuse in the opinion of the investigator.
4. Any disease or condition, physical or psychological that, in the opinion of the investigator, would compromise the safety of the subject or the likelihood of achieving reliable results or increase the likelihood of the subject being withdrawn.
5. Laboratory findings at screening which, in the opinion of the investigator, are clinically significant for this subject population.
6. A screen serum magnesium concentration of >1.25 mmol/L (>3.0 mg/dL).
7. A known history of haemochromatosis.
8. Subjects receiving either tetracycline or lithium treatment.
9. A serum ferritin level of ≥1000 ng/mL.
10. Non-elective hospitalisation in the 4 weeks prior to screening.
11. Female subjects who are of childbearing potential and who are neither surgically sterilised nor using reliable contraceptive methods (hormonal, barrier methods or intrauterine device) or who are lactating or pregnant.
12. Current hypophosphataemia at screening (last 2 consecutive phosphate values of <0.7 mmol/L [<2.2 mg/dL]).
13. Known history of colorectal malignancy, familial polyposis coli and/or strong family history (in 2 or more first degree relatives) of these terms.
14. A QTcF interval of >560 ms at screen.
15. Known persistent (>1 month) non compliance (<70%) with prescribed medication regimens at screen.
16. Current clinically significant intestinal motility disorder.
17. Bowel obstruction with current or previous use of sevelamer HCl.
18. Known intolerance to sevelamer HCl or any excipients of fermagate or Renagel medication.
19. Subjects with inflammatory bowel disease that, in the investigator's opinion, is poorly controlled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Control or not the level of serum phosphate | Within the treatment period

SECONDARY OUTCOMES:
Change from baseline in mean serum phosphate | End of 3 months treatment in maintenance period
Change from baseline in calcium, calcium phosphate product and PTH level | End of 3 months treatment in maintenance period

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer (Information at Ineos Healthcare Limited), Dr., Study Chair — Ineos Healthcare Limited
Locations (109):
- United States (40):
  - Arkansas Nephrology Services Ltd, Hot Springs, Arkansas
  - National Institute of Clinical Research, Bakersfield, California
  - Renal Medical Associates, Lynwood, California
  - Academic Medical Research Institute Inc, Monterey Park, California
  - Pasadena Nephrology, Pasadena, California
  - Sierra View Nephrology SC, Porterville, California
  - Kidney Center Inc., Thousand Oaks, California
  - Stanford Nephrology, Stamford, Connecticut
  - Capitol Dialysis, Washington D.C., District of Columbia
  - Discovery Medical Research Group Inc., Ocala, Florida
  - Cleveland William MD, Atlanta, Georgia
  - Davita South Brunswick Dialysis Center, Brunswick, Georgia
  - North Shore University Health System, Evanston, Illinois
  - Southwest Nephrology Associates, Evergreen Park, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Renal Associates of Baton Rouge, Baton Rouge, Louisiana
  - Western New England Transplant Associates, Springfield, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Huq Cruz Strauss Masud PA, Neptune City, New Jersey
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Nassau Nephrology, LLP, Bellmore, New York
  - Clinical Research Development Associates LLC, Springfield Gardens, New York
  - Nephrology Associates, PA, Winston-Salem, North Carolina
  - Bayview Nephrology, Erie, Pennsylvania
  - Renal Endocrine Associates PC, Pittsburgh, Pennsylvania
  - Renal-Endocrine Associates, Pittsburgh, Pennsylvania
  - CSRA Renal Services, Aiken, South Carolina
  - Carolina Diabetes & Kidney Center, Sumter, South Carolina
  - Carolina Diabetes and Kidney Center/ sumter Medical Specialist, Sumter, South Carolina
  - South Arlington Dialysis Center, Arlington, Texas
  - U.S Renal Care, Grand Prairie, Texas
  - U.S. Renal Care, Grand Prairie, Texas
  - Diagnostic Clinic of Houston, Houston, Texas
  - SouthWest Houston Research LTD., Houston, Texas
  - Renal Associates PA, San Antonio, Texas
  - University of Vermont, Burlington, Vermont
  - Ramon Mendez MD PC (private practice), Alexandria, Virginia
  - Ramon Mendez, MD, PC (private practice), Alexandria, Virginia
  - Clinical Research & Consulting Center LLC, Fairfax, Virginia
- Belgium (5):
  - O.L.V Ziekenhuis, Aalst
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Brussel, Jette
  - U. Z. Gasthuisberg, Leuven
  - Hôpital de la Citadelle, Liège
- Brazil (3):
  - Nefroclinica de Uberlandia Ltda, Uberlândia, Minas Gerais
  - Hospital Geral de Bonsucesso, Rio de Janeiro, Rio de Janeiro
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
- Bulgaria (11):
  - MHAT - Pazardzhik AD, Pazardzhik
  - University Multiprofile Hospital for Active Treatment "Dr. G. Stransky", Pleven
  - MHAT - Plovdiv AD, Plovdiv
  - MHAT - Rousse AD, Rousse
  - MHAT 'Tokuda Hospital Sofia' AD, Sofia
  - UMHAT 'Alexandrovska', Sofia
  - UMHAT 'Sv. Ivan Rilski' EAD, Sofia
  - Multiprofile Hospital for Active Treatment and Emergency Medicine "Pirogov", Sofia
  - MHAT 'Sv. Anna - Varna' AD, Varna
  - MHAT 'Sveta Marina', Varna
  - Centre of Haemodialysis and Nephrology MHAT 'Dr. Stefan Cherkezov' AD, Veliko Tarnovo
- Czechia (6):
  - Fakultní nemocnice u sv. Anny, Brno
  - Krajska nemocnice Liberec, a.s., Liberec
  - Nemocnice v Prachaticich, a.s., Prachatice
  - VFN Praha, Prague
  - Nemocnice Tabor a.s., Tábor
  - Nemocnice Znojmo, Znojmo
- Estonia (3):
  - West-Tallinn Central Hospital, Tallinn
  - North Estonia Regional Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Hungary (4):
  - FMC Dialysis Centre, Budapest
  - Diaverum Dialysis Centre, Hódmezővásárhely
  - FMC Dializis Center Kecskemet, Kecskemét
  - FMC Dializis Centrum Kft Vac Javorszky Odon Korhaz, Vác
- Israel (3):
  - Barzilai Medical Center, Ashkelon
  - Assaf Harofeh Medical Center, Beer Yaakov
  - Western Galilee Hospital - Nahariya, Nahariya
- Italy (3):
  - Azienda Ospedaliera Istituti Ospitalieri di Cremona, Cremona, CR
  - Azienda Ospedaliera Policlinico di Modena, Modena, MO
  - Fondazione "S. Maugeri" IRCCS, Pavia, PV
- Lithuania (8):
  - Diaverum klinikos JSC, Kaunas
  - Kaunas Medical University Hospital Public Institution, Kaunas
  - B.Braun Avitum JSC, Kaunas
  - Diaverum klinikos JSC, Kėdainiai
  - Diaverum klinikos JSC, Klaipėda
  - Siauliai Regional Hospital Public Institution, Šiauliai
  - Diaverum klinikos JSC, Vilnius
  - Vilnius City University Hospital Public Institution, Vilnius
- Hospital y Clinica OCA SA de CV, Monterrey, Mexico
- Serbia (4):
  - Clinical Center Zvezdara, Belgrade
  - Clinical Center Nis, Niš
  - Clinical Centre of Vojvodina, Novi Sad
  - Clinical Center Zemun, Zemun
- Slovakia (4):
  - Logman a.s., Banská Bystrica
  - Nephro s.r.o. Levice, Levice
  - Privat Nephro-Dialysis Centre Ldt Martin, Martin
  - LOGMAN a.s., Trenčín
- South Africa (5):
  - N1 City Hospital, Cape Town, Western Cape
  - South Peninsula Dialysis, Cape Town, Western Cape
  - Grootte Schuur Hospital, Cape Town, Western Cape
  - Panorama Medi Clinic, Parow, Western Cape
  - Tygerberg Hospital, Parow, Western Cape
- United Kingdom (9):
  - Addenbrooke's Hospital, Cambridge, Cambs
  - The Royal London Hospital, London, Gt Lon
  - Leicester General Hospital, Leicester, Leics
  - Royal Liverpool Hospital, Liverpool, Mersyd
  - Norfolk and Norwich University Hospital, Norwich, Norflk
  - St Lukes Hospital, Bradford, Nthumb
  - University Hospital of Wales, Cardiff, S Glam
  - Royal Berkshire Hospital, Reading
  - Northern General Hospital, Sheffield